CLINICAL TRIAL: NCT04300218
Title: Effectiveness and Cost-effectiveness of iCBT-I in Clinical Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Collaborators: University of Bern (Other)
Responsible Party: Principal Investigator, Poluektov Mikhail Gur'evich, Assoc.prof, Dr., I.M. Sechenov First Moscow State Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 03-20
Record Dates: First submitted 2020-03-03; First posted 2020-03-09 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Chronic Insomnia
Keywords: cognitive-behavioral psychotherapy; online Intervention; cost-effectiveness; chronic insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Multicenter parallel-group add-on superiority randomized controlled trial (RCT) comparing an active treatment condition (iCBT-I plus CAU) to CAU alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCBT-I + CAU (Experimental): Participants of this arm will get access to the course of the online cognitive-behavioral therapy for insomnia (iCBT-I) for 2 months along with the treatment prescribed by a consulting doctor (care as usual - CAU). After the 2-month course participants will pass the post-treatment assessment followed by the 3-month follow-up and post-follow-up assessment
  Interventions: Behavioral: internet-delivered cognitive-behavioral therapy for insomnia (iCBT-I); Other: Care as usual (CAU)
- CAU (Active Comparator): Participants of this arm will get a treatment prescribed by a consulting doctor (care as usual - CAU). After the 2-month course participants will pass the post-treatment assessment followed by the 3-month follow-up and post-follow-up assessment. Then provided completion of all the assessments and satisfying eligibility criteria participants of this arm will get tha access to the 2-month iCBT-I course followed by the post-treatment assessment
  Interventions: Behavioral: internet-delivered cognitive-behavioral therapy for insomnia (iCBT-I); Other: Care as usual (CAU)

INTERVENTIONS:
Behavioral: internet-delivered cognitive-behavioral therapy for insomnia (iCBT-I) — The 2-month intervention consists of educational material divided into 8 modules, which provide the rationale for the CBT-I interventions: sleep restriction; stimulus control; cognitive techniques; relaxation techniques. Information is presented in 10-minute videolectures.
  The program includes a sleep diary to insert bedtime and waketime, sleep latency, total sleep time, night awakenings.
  All material will be delivered through the internet program and expected to be elaborated by the patient but with the opportunity to contact a specialist via the feedback form (guidance on request) in a secured environment if they face difficulties or possible negative effects of the intervention. The content of the program is based on an already established internet-based self-help program against insomnia that was already tested in a previous study.
Other: Care as usual (CAU) — Intervention includes all variety of therapy methods that can be prescribed by medical doctors (MD): pharmacotherapy, behavioral recommendations, face-to-face psychotherapy. Prescriptions may be made during the first visit to MD, or at any point in the study on a next doctor visit, or during visits to the doctors of other medical centers. All concurrently applied treatments will be assessed repeatedly by self-report

SUMMARY:
The proposed parallel-group randomized controlled trial add-on superiority of the iCBT-I program with CAU as a control condition will let us investigate the effectiveness and cost-effectiveness of iCBT-I. Analysis of baseline characteristics of the participants aims to find predictors of outcome

DETAILED DESCRIPTION:
Application of internet-delivered cognitive-behavior treatment for insomnia (iCBT-I) is a perspective method that can fill the gap created by the discrepancy between insomnia cases and the number of trained professionals. Although the effectiveness of this method was proven in multiple studies conducted in research settings, it is unclear if iCBT-I outperforms pharmacotherapy which remains a widely used alternative of cognitive-behavior therapy of insomnia (CBT-I). Predictors, mediators, and moderators of treatment effect remain uncertain since previous studies often give contradictory results. The present study aims to investigate clinical effectiveness and cost-effectiveness of an internet-based CBT-I program Sleepsy in comparison with care as usual (CAU) among patients with chronic insomnia (CI) recruited from clinical settings. Baseline data will be further analyzed to find predictors of treatment outcome

For these purposes, a parallel-group randomized controlled trial add-on superiority of the iCBT-I program with CAU as a control condition was designed. 110 participants will be referred from the medical doctors in Moscow. Both groups will have access to CAU, treatment prescribed by the referred doctor. Patients of the first group will additionally get access to the iCBT-I program with the opportunity to contact a specialist within the program (guidance on request) in a secured environment. The primary outcome is insomnia severity change from pre- to posttreatment and to post-follow-up. Secondary outcomes include change subjective sleep characteristics, daytime symptoms, comorbid affective disorders, dysfunctional cognitions and behavior, healthcare consumption, and productivity losses. Predictors analysis will include baseline scores of the aforementioned outcomes along with treatment expectancies, personality traits

To the best of our knowledge, the present study is the first study of iCBT-I to be conducted in clinical settings. We expect that this approach lets us determine the target group more precisely and exclude health problems that may interfere with treatment. It is also expected that patients, referred to iCBT-I from the doctor's office will be more motivated to finish the treatment course that will reduce the drop out rate. CAU as control condition let us reconstruct clinical situation facing practicing doctor. On the other hand, CAU may result in a loss of power to detect a meaningful difference. Limitation of our study is in the impossibility of blinding participants to the treatment condition

ELIGIBILITY:
Inclusion Criteria:

* Sleep disorder matching chronic insomnia criteria (International Classification of Sleep Disorders-3) - assessed by clinical judgement
* Ability to follow the procedures of the study, fluent Russian language, Good access to internet - assessed by self-report

Exclusion Criteria:

* Presence of dementia (identified by history or a score < 25 on the Folstein Mini Mental Status Exam) - assessed by clinical judgement
* Severe depression or severe anxiety as measured with the Beck Depression Inventory (BDI-II; score > 28 ) and the Beck Anxiety Inventory (BAI; score > 26) - assessed by the questionnaires
* History of severe psychiatric comorbidities other than anxiety and depression (bipolar disorders, psychotic disorders) or substance use disorder - assessed by self-report and clinical history
* Untreated severe obstructive sleep apnea syndrome (apnea-hypopnea index (AHI) > 15), restless legs syndrome (movement index with arousal > 15 per hour) or other sleep disorders affecting night sleep - assessed by clinical judgement and clinical history
* pregnancy, lactation - assessed by self-report
* having a serious somatic condition or brain disorders (stroke, Parkinson's disease…) preventing further participation - assessed by self-report
* Having high suicidality risk - assessed by clinical judgement, high total BDI-II score (> 29) or score >1 on a BDI-II of suicidality subscale

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail G Poluektov, PhD, Principal Investigator — I.M.Sechenov First Moscow Medical University
Locations (3):
- Russia (3):
  - Sleep medicine department, University clinical hospital 3, I.M.Sechenov First Moscow Medical University, Moscow, Moscow
  - Stavropol regional somnological center, Stavropol, Stavropol Kray
  - Kuzbass clinical veterans hospital, Kemerovo

IPD SHARING:
Plan to Share IPD: Yes
Results of this trial will be disseminated via peer-reviewed journal publications. Primary and secondary aims will be reported in a single publication. Other findings will be published separately. T
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Pchelina P, Poluektov M. Duration of insomnia and success expectancy predict treatment outcome of iCBT for insomnia. Front Sleep. 2024 Nov 6;3:1415077. doi: 10.3389/frsle.2024.1415077. eCollection 2024. PMID 41424507
- [Derived] Pchelina P, Poluektov M, Krieger T, Duss SB, Berger T. Clinical effectiveness of internet-based cognitive behavioral therapy for insomnia in routine secondary care: results of a randomized controlled trial. Front Psychiatry. 2024 May 10;15:1301489. doi: 10.3389/fpsyt.2024.1301489. eCollection 2024. PMID 38800061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 115 patients with chronic insomnia fulfilling ICSD-3 criteria referred from neurologists specialized in somnology in Moscow (Sleep Medicine department, University Clinic 3, Sechenov First Moscow State Medical University, Moscow) from March 2020 to December 2022 were assessed for eligibility
Groups:
- iCBT-I + CAU: Participants of this arm will get access to the course of the online cognitive-behavioral therapy for insomnia (iCBT-I) for 2 months along with the treatment prescribed by a consulting doctor (care as usual - CAU).
  The 2-month intervention consists of educational material divided into 8 modules, which provide the rationale for the CBT-I interventions: sleep restriction; stimulus control; cognitive techniques; relaxation techniques. Information is presented in 10-minute videolectures.
  The program includes a sleep diary to insert bedtime and waketime, sleep latency, total sleep time, night awakenings.
  All material will be delivered through the internet program and expected to be elaborated by the patient but with the opportunity to contact a specialist via the feedback form (guidance on request) in a secured environment if they face difficulties or possible negative effects of the intervention. The content of the program is based on an already established internet-based self-help program against insomnia that was already tested in a previous study.
  Care as usual (CAU): Intervention includes all variety of therapy methods that can be prescribed by medical doctors (MD): pharmacotherapy, behavioral recommendations, face-to-face psychotherapy. Prescriptions may be made during the first visit to MD, or at any point in the study on a next doctor visit, or during visits to the doctors of other medical centers.
- Care as Usual (CAU): Participants of this arm will get a treatment prescribed by a consulting doctor (care as usual - CAU).
  Care as usual (CAU): Intervention includes all variety of therapy methods that can be prescribed by medical doctors (MD): pharmacotherapy, behavioral recommendations, face-to-face psychotherapy. Prescriptions may be made during the first visit to MD, or at any point in the study on a next doctor visit, or during visits to the doctors of other medical centers. All concurrently applied treatments will be assessed repeatedly by self-report
Period: Overall Study
Arm/Group | iCBT-I + CAU | Care as Usual (CAU)
Started | 53 | 54
Completed | 47 | 46
Not Completed | 6 | 8
Not completed — Lost to Follow-up | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- iCBT-I + CAU: Demographic characteristics and baseline clinical scores for the study sample were compared with t-test and Chi-square test. iCBT-I + CAU group participants were significantly younger:median (IQR) = 37 (28-50); and had lower FSS: mead (SD) = 36.2 (15.4) Medications used for the management of insomnia included benzodiazepines and hypnotic benzodiazepine receptor agonists, sedating antidepressants, antipsychotics, antihistamines, melatonin, phytotherapy, and off-label substances
- Care as Usual (CAU): Demographic characteristics and baseline clinical scores for the study sample were compared with t-test and Chi-square test. iCBT-I + CAU group participants were significantly older: median (IQR) = 40.5 (34.2-60.5); and had higher FSS: mead (SD) = 43.2 (12.4). Medications used for the management of insomnia included benzodiazepines and hypnotic benzodiazepine receptor agonists, sedating antidepressants, antipsychotics, antihistamines, melatonin, phytotherapy, and off-label substances.
- Total: Total of all reporting groups
Arm/Group | iCBT-I + CAU | Care as Usual (CAU) | Total
Number analyzed (Participants) | 53 | 54 | 107
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [28 to 50] | 40.5 [34.2 to 60.5] | 40 [31.5 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 62
  Male | 23 | 22 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 53 | 54 | 107
ISI - insomnia severity index [Mean (Standard Deviation); unit: units on a scale] — is a seven-item insomnia assessment tool. The 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28 where higher score reflects more severe insomnia. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28)
  units on a scale | 15.4 (4.2) | 15.4 (3.9) | 15.4 (4.0)
BDI - Beck depression inventory [Mean (Standard Deviation); unit: units on a scale] — 21-question with a 4-point Likert scale and ranging answers from 0 to 3, yielding a total score ranging from 0 to 63 with higher score reflecting more severe depression. A BDI cutoff higher than 28 indicates severe depression.
  units on a scale | 10.7 (5.7) | 12.4 (6.5) | 11.6 (6.2)
BAI - Beck anxiety inventory [Mean (Standard Deviation); unit: units on a scale] — 21-question inventory with a 4-point Likert scale and ranging answers from 0 to 3, yielding a total score ranging from 0 to 63 with higher score reflecting more severe anxiety. A BDI cutoff higher than 28 indicates severe depression.
  units on a scale | 8.7 (6.9) | 10.3 (7.4) | 9.5 (7.1)
SF-12 - quality of life short-form survey [Mean (Standard Deviation); unit: units on a scale] — The 12-item Short Form Survey (SF-12) contains categorical questions (yes/no) and questions with a 3, 5 and 6-point Likert scale. The SF-12 total score is a summary of mental health (MCS12), and physical health (PCS12). Scores range from 0 to 100, with higher scores indicating better functioning. The scores are represented as T-scores that are linear transformations with a mean of 50 and a standard deviation of 10 in the general population. A score of < 50 on the PCS-12 is a cut-off to determine a physical condition; score of <42 on the MCS-12 may be indicative of 'clinical depression'
  units on a scale | 31.7 (5.6) | 31.1 (5.5) | 31.4 (5.6)
FSS - fatigue severity scale [Mean (Standard Deviation); unit: units on a scale] — Consists of 9 items with 7-point Likert scale (from 1 to 7). The minimum total score=9 and maximum score possible=63. Higher total score corresponds to greater fatigue severity. A total score of less than 36 suggests that the subject may not be suffering from fatigue
  units on a scale | 36.2 (15.4) | 43.2 (12.4) | 39.8 (14.3)
ESS - epworth sleepiness scale [Mean (Standard Deviation); unit: units on a scale] — a measure asking propensity for "dosing" in eight daytime situations on the 4/point Likert scale from 0 = never to 3= very high propensity, yielding a total score ranging from 0 (no sleepiness) to 24 (high sleepiness), with normal score < 9.
  units on a scale | 4.8 (4.1) | 5.5 (3.9) | 5.2 (4.0)
DBAS - dysfunctional beliefs about sleep scale [Mean (Standard Deviation); unit: units on a scale] — The questionnaire consists of 16 questions with a Likert scale ranging answers from 0 = strongly disagree to 10 = strongly agree with a total score ranging from 0 to 160. Higher total score reflects more prominent dysfunctional beliefs about sleep. The scale has no cutoff score
  units on a scale | 101.2 (25.8) | 109.8 (22.5) | 105.6 (24.5)
LCS - locus control of sleep scale [Mean (Standard Deviation); unit: units on a scale] — Measure Description: The questionnaire consists of 8 questions with a Likert scale ranging answers from 1 = strongly disagree to 6 = strongly agree with a total score ranging from 8 to 48 with higher scores reflecting a more internal sleep locus of control. The scale has no cutoff score
  units on a scale | 42.2 (11.8) | 41.7 (14.0) | 42.0 (12.9)
SHI - sleep hygiene index [Mean (Standard Deviation); unit: units on a scale] — A 13-question questionnaire evaluating each item on a 5-point Likert scale from 1 to 5, yielding a total score ranging from 13 to 65. Higher total score reflects worse sleep hygiene. The questionnaire has no cutoff score
  units on a scale | 47.7 (8.2) | 47.5 (6.8) | 47.6 (7.5)
SE - sleep effectiveness [Mean (Standard Deviation); unit: percentage of time in bed spent asleep] — subjective sleep measure calculated as the ratio between the total sleep time, and the time spent in bed. Both total sleep time and time spent in bed are derived from the sleep diary. For the study we used the mean sleep efficiency for one week
  percentage of time in bed spent asleep | 75.4 (12.8) | 78.9 (11.1) | 77.2 (12.1)
SOL - sleep onset latency [Mean (Standard Deviation); unit: minutes] | 40.7 (28.7) | 45.2 (39.6) | 43.0 (34.6)
WASO - wake after sleep onset [Mean (Standard Deviation); unit: minutes] | 40.5 (43.3) | 32.6 (35.2) | 36.5 (39.4)
TST - total sleep time [Mean (Standard Deviation); unit: hours] | 6.7 (1.6) | 6.8 (1.6) | 6.7 (1.4)
Duration of insomnia [Median (Inter-Quartile Range); unit: months] | 36 [18 to 66.5] | 48 [12 to 84] | 36 [17.75 to 79.5]
Use of medications for insomnia, n (%) [Count of Participants; unit: Participants] | 47 | 42 | 89
Use of benzodiazepines and/or Z-drugs for insomnia, n (%) [Count of Participants; unit: Participants] — This measure was collected by a question if the subject was ever prescribed medications for insomnia treatment. If the subject replied yes, they were requested to fill in the name, dose and duration of use of the medication. Further, the answers were manually transformed into the categorical (yes or no) variable reflecting the use of benzodiazepines and/or Z-drugs (zopiclone, zolpidem, zaleplon)
  Participants | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (ISI)
Description: Change of ISI from pre- to post-treatment and post-follow-up. Change is calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the better outcome, negative values correspond to the worse outcome, i.e. increase of insomnia severity.
  The ISI is a seven-item insomnia assessment tool. The 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28)
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- iCBT-I + CAU: Participants of this arm will get access to the course of the online cognitive-behavioral therapy for insomnia (iCBT-I) for 2 months along with the treatment prescribed by a consulting doctor (care as usual - CAU).
  internet-delivered cognitive-behavioral therapy for insomnia (iCBT-I): The 2-month intervention consists of educational material divided into 8 modules, which provide the rationale for the CBT-I interventions: sleep restriction; stimulus control; cognitive techniques; relaxation techniques. Information is presented in 10-minute videolectures. The program includes a sleep diary to insert bedtime and waketime, sleep latency, total sleep time, night awakenings. All material will be delivered through the internet program and expected to be elaborated by the patient but with the opportunity to contact a specialist via the feedback form (guidance on request) in a secured environment if they face difficulties or possible negative effects of the intervention. The content of the program is based on an already established internet-based self-help program against insomnia that was already tested in a previous study.
  Care as usual (CAU): Intervention includes all variety of therapy methods that can be prescribed by medical doctors (MD): pharmacotherapy, behavioral recommendations, face-to-face psychotherapy. Prescriptions may be made during the first visit to MD, or at any point in the study on a next doctor visit, or during visits to the doctors of other medical centers.
- Care as usual (CAU): Participants of this arm will get a treatment prescribed by a consulting doctor (care as usual - CAU). After the 2-month course participants will pass the post-treatment assessment followed by the 3-month follow-up and post-follow-up assessment. Then provided completion of all the assessments and satisfying eligibility criteria participants of this arm will get tha access to the 2-month iCBT-I course followed by the post-treatment assessment Care as usual (CAU): Intervention includes all variety of therapy methods that can be prescribed by medical doctors (MD): pharmacotherapy, behavioral recommendations, face-to-face psychotherapy. Prescriptions may be made during the first visit to MD, or at any point in the study on a next doctor visit, or during visits to the doctors of other medical centers.
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale
  change from pre- to post-treatment | 10.0 (5.1) | 13.5 (5.5)
  change from pre-treatment to follow-up | 11.3 (5.7) | 13.1 (5.7)

2. Secondary Outcome: Sleep Onset Latency (SOL),
Description: Sleep diary derived measure averaged for 1 week pre- post-treatment, post-follow-up. For the purposes of effectiveness investigation change of SOL from pre- to post-treatment and post-follow-up. Change of SOL is calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the better outcome, negative values correspond to the worse outcome, i.e. increase of sleep latency
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Median (Standard Deviation); unit: minutes
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
minutes
  change from pre- to post-treatment | 28.2 (29.0) | 39.2 (37.2)
  change from pre-treatment to follow-up | 33.3 (28.2) | 42.5 (37.1)

3. Secondary Outcome: Total Sleep Time (TST)
Description: Sleep diary derived measure averaged for 1 week pre- post-treatment, post-follow-up. For the purposes of effectiveness investigation change of TST from pre- to post-treatment and post-follow-up. Change of TST is calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the worse outcome, negative values correspond to the better outcome, i.e. increase of total sleep time
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
hours
  pre- to post-treatment change | 6.9 (1.3) | 7.0 (1.2)
  change from pre-treatment to follow-up | 7.3 (1.3) | 7.0 (1.1)

4. Secondary Outcome: Sleep Efficiency (SE)
Description: Sleep diary derived measure calculated as the ratio of TST to time spent in bed multiplied by 100%, averaged for 1 week pre- post-treatment, post-follow-up. For the purposes of effectiveness investigation change of SOL from pre- to post-treatment and post-follow-up. Change of SE is calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the worse outcome, negative values correspond to the better outcome, i.e. increase of sleep efficiency
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
percent
  change pre- to post-treatment | 84.5 (10.4) | 81.9 (9.9)
  change from pre-treatment to follow-up | 83.8 (8.2) | 80.2 (11.9)

5. Secondary Outcome: Wake After Sleep Onset (WASO)
Description: Sleep diary derived measure averaged for 1 week pre- post-treatment, post-follow-up. For the purposes of effectiveness investigation change of WASO from pre- to post-treatment and post-follow-up. Change of WASO is calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the better outcome, negative values correspond to the worse outcome, i.e. increase of the time spent awake after sleep onset
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
minutes
  change pre- to post-treatment | 19.0 (16.7) | 28.0 (35.2)
  change pre-treatment to follow-up | 28.8 (22.0) | 29.3 (29.3)

6. Secondary Outcome: Fatigue Severity Scale (FSS)
Description: Disorder non-specific 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle. Each item is evaluated on the 7 points Likert scale (e.g., 1 indicates strongly disagree and 7=strongly agree.), yielding a total score ranging from 9 to 63. A higher score reflects a higher level of fatigue. Change of FSS was calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the better outcome, negative values correspond to the worse outcome, i.e. increase of fatigue
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale
  change from pre- to post-treatment | 35.1 (14.0) | 40.6 (13.8)
  change from pre-treatment to follow-up | 33.3 (14.9) | 38.3 (15.2)

7. Secondary Outcome: Short-form Survey (SF-12 Version 1.0)
Description: The Short Form Survey (SF-12)is calculated as a summary of the mental component score (MCS-12) and a physical component score (PCS-12). Total score ranges from 0 to 100, with higher scores indicating better functioning. The subscale scores are represented as T-scores with a mean of 50 and a standard deviation of 10 in the general population. A score of < 50 on the PCS-12 is a cut-off to determine a physical condition; score of <42 on the MCS-12 may be indicative of 'clinical depression'. For this study we used change of the SF-12 total score as outcome. Change of SF-12 is calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the worse outcome, negative values correspond to the better outcome, i.e. increase of physical and mental health functioning
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale
  change pre- to post-treatment | 34.7 (5.6) | 33.1 (6.3)
  change from pre-treatment to follow-up | 33.7 (6.6) | 32.8 (6.2)

8. Secondary Outcome: Epworth Sleepiness Scale (ESS)
Description: Measure asking propensity for 'dosing' in eight daytime situations from 0 = never to 3= very high propensity, yielding a total score ranging from 0 to 24 with normal score < 9. Change of ESS is calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the better outcome, negative values correspond to the worse outcome, i.e. increase of daytime sleepiness
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale
  change from pre- to post-treatment | 4.4 (3.9) | 4.1 (3.6)
  change from pre-treatment to follow-up | 3.9 (4.5) | 4.0 (2.9)

9. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: 21-questions inventory with a 4-point Likert scale and ranging answers from 0 to 3, yielding a total score ranging from 0 to 63. A BAI total score higher than 25 corresponds to severe anxiety. Change of BAI is calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the better outcome, negative values correspond to the worse outcome, i.e. increase of anxiety
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale
  Change from pre- to post-treatment | 7.0 (6.4) | 9.8 (7.7)
  Change from pre-treatment to follow-up | 8.3 (7.9) | 9.3 (7.6)

10. Secondary Outcome: Beck Depression Inventory (BDI-II)
Description: 1-questions inventory with a 4-point Likert scale and ranging answers from 0 to 3, yielding a total score ranging from 0 to 63. A BDI cutoff higher than 28 indicates severe depression. Change of BDI-II is calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the better outcome, negative values correspond to the worse outcome, i.e. increase of depression
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale
  Change from pre- to post-treatment | 6.7 (5.2) | 10.2 (5.4)
  Change from pre-treatment to follow-up | 8.0 (6.2) | 10.3 (7.0)

11. Secondary Outcome: Sleep Hygiene Index (SHI)
Description: 13-questions questionnaire evaluating each item on a 5-point Likert scale, yielding a total score ranging from 13 to 65. Higher SHI score corresponds to the worse sleep hygiene. Change of SHI is calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the better outcome, negative values correspond to the worse outcome, i.e. worsening of sleep hygiene habits
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale
  change from pre- to post-treatment | 51.9 (7.2) | 49.8 (6.5)
  change from pre-treatment to follow-up | 27.7 (7.7) | 28.5 (6.3)

12. Secondary Outcome: Sleep Locus of Control Questionnaire (SLC)
Description: variant validated in Russia comprises 8 questions scored using a 6-point Likert scale ranging each answer from 1 = strongly disagree; 6 = strongly agree, yielding a total score ranging from 8 to 48. The Russian adaptation of the scale has shown internal reliability of 0.41. Higher SLC score corresponds to the more marked external locus of control. Change of SLC is calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the better outcome, negative values correspond to the worse outcome, i.e. more prominent external locus of control of sleep
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale
  change from pre- to post-treatment | 38.5 (9.6) | 38.6 (9.9)
  change from pre-treatment to folow-up | 39.8 (12.0) | 40.1 (13.6)

13. Secondary Outcome: Dysfunctional Beliefs and Attitudes About Sleep Scale (DBAS)
Description: designed to identify and assess the severity of various sleep and insomnia-related cognitions. It consists of 16 questions with a Likert scale ranging answers from 0 = strongly disagree to 10 = strongly agree with a total score ranging from 0 to 160. Higher DBAS score reflects more severe dysfunctional thinking. The Russian adaptation of the scale has high internal reliability of 0.86. Change of DBAS is calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the better outcome, negative values correspond to the worse outcome, i.e. more prominent dysfunctional beliefs about sleep
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale
  change from pre- to post-treatment | 75.3 (31.5) | 95.8 (27.2)
  change from pre-treatment to follow-up | 76.1 (33.6) | 99.3 (27.7)

14. Secondary Outcome: Anxiousness Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Anxiousness is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- CAU group: Participants of this arm will get a treatment prescribed by a consulting doctor (care as usual - CAU).
  Care as usual (CAU): Intervention includes all variety of therapy methods that can be prescribed by medical doctors (MD): pharmacotherapy, behavioral recommendations, face-to-face psychotherapy. Prescriptions may be made during the first visit to MD, or at any point in the study on a next doctor visit, or during visits to the doctors of other medical centers. All concurrently applied treatments will be assessed repeatedly by self-report
Arm/Group | iCBT-I + CAU | CAU group
Number analyzed (Participants) | 53 | 54
score on a scale | 2.43 (0.84) | 2.62 (0.75)

15. Secondary Outcome: Trimbos Questionnaire for Costs Associated With Psychiatric Illness (TiC-P) Health Care Consumption
Description: This measure aims to evaluate the cost-effectiveness of iCBT-I. The first part of TIC-P consists of 14 questions on the volume of health care uptake: including the number of medical consultations, dose, and frequency of medication, days of inpatient care. Multiplication of these data by the actual price of medical help produces the cost of medical care as the outcome. The higher outcome represents higher costs of medical care. Change of TiC-P Health care consumption is calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the better outcome, negative values correspond to the worse outcome, i.e. higher costs of the healthcare consumption
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Median (Inter-Quartile Range); unit: roubles
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
roubles
  Change from pre- to post-treatment | 16500 [12100 to 26818] | 4896 [0 to 9340]
  Change from pre-treatment to follow-up | 6263 [790 to 16630] | 5959 [1333 to 10097]

16. Secondary Outcome: Trimbos Questionnaire for Costs Associated With Psychiatric Illness (TiC-P) Short Form- Health and Labour Questionnaire (SF-HLQ)
Description: This measure aims to evaluate the cost-effectiveness of iCBT-I. The second part of TIC-P is represented by the Short Form- Health and Labour Questionnaire (SF-HLQ), an instrument to collect data on productivity losses (presenteeism and absenteeism) due to health problems. Costs of productivity losses are calculated by multiplication of missed working hours by standard cost price of productivity. The higher outcome represents higher costs of productivity losses. Change of TiC-P productivity losses is calculated as the value at the earlier time point minus the value at the later time point. Positive values correspond to the better outcome, negative values correspond to the worse outcome, i.e. higher costs of the productivity losses
Time Frame: pre- to post-treatment 2 months, pre-treatment to follow-up 5 months
Measure: Median (Inter-Quartile Range); unit: roubles
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
roubles
  Change from pre- to post-treatment | 2449 [0 to 17975] | 7238 [0 to 14694]
  Change from pre-treatment to follow-up | 1196 [0 to 7698] | 2853 [396 to 8002]

17. Secondary Outcome: Success Expectancy
Description: Aims to measure patients' beliefs about the expected treatment success as one of the important outcome predictors. For its evaluation we will use one adapted question of Credibility/Expectancy Questionnaire: "At this point, how successfully do you think this treatment will be in reducing your insomnia symptoms?" at scale from 1 to 9. This question was chosen as well representing high correlation for both factors: credibility and expectancy, and most logically formulated for the intended purpose
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Care as usual (CAU): Care as usual (CAU): Intervention includes all variety of therapy methods that can be prescribed by medical doctors (MD): pharmacotherapy, behavioral recommendations, face-to-face psychotherapy. Prescriptions may be made during the first visit to MD, or at any point in the study on a next doctor visit, or during visits to the doctors of other medical centers.
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
score on a scale | 6.3 (1.57) | 6.2 (1.64)

18. Secondary Outcome: User Satisfaction
Description: feedback questionnaire developed for this study. It includes 1 question about satisfaction or dissatisfaction with the treatment with a 5-point Likert scale, from 1 (very poor/not at all useful) to 5 (very, good/very useful).
  The questionnaire also contains open questions aiming for utilitarian goals, i.e. to improve the program (possible negative effects of the intervention if any: deterioration of insomnia symptoms, adverse effects, novel symptoms; and about improvement suggestions, what participants liked most if they would recommend it to a friend with insomnia). These questions are not included in questionnaire score
Time Frame: After completion of iCBT-I course: week 8 after randomization for arm iCBT-I +CAU; week 28 after randomization for arm CAU
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 1
score on a scale | 3.7 (1.28) | 5.0 (NA) — Only 1 participant of CAU group replied this question

19. Secondary Outcome: System Usability Scale (SUS)
Description: 10-item non-specific questionnaire used to collect a user's subjective rating of a product's (products, websites, applications, hardware, or software) usability and learnability. Each item is scored on a scale of 0 ("strongly Disagree") to 4 ("strongly Agree"). For positively-worded items (1, 3, 5, 7 and 9), the score contribution is the scale position minus 1. For negatively-worded items (2, 4, 6, 8 and 10), it is 5 minus the scale position. To get the overall SUS score, multiply the sum of the item score contributions by 2.5. Thus, SUS scores range from 0 to 100 in 2.5-point increments. Higher SUS score reflects better subjective usability of the program.
Time Frame: as for outcome 18
Population: data were not analyzed
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- iCBT-I + CAU: Participants of this arm will get access to the course of the online cognitive-behavioral therapy for insomnia (iCBT-I) for 2 months along with the treatment prescribed by a consulting doctor (care as usual - CAU). After the 2-month course participants will pass the post-treatment assessment followed by the 3-month follow-up and post-follow-up assessment
  internet-delivered cognitive-behavioral therapy for insomnia (iCBT-I): The 2-month intervention consists of educational material divided into 8 modules, which provide the rationale for the CBT-I interventions: sleep restriction; stimulus control; cognitive techniques; relaxation techniques. Information is presented in 10-minute videolectures.
  The program includes a sleep diary to insert bedtime and waketime, sleep latency, total sleep time, night awakenings.
  All material will be delivered through the internet program and expected to be elaborated by the patient but with the opportunity to contact a specialist via the feedback form (guidance on request) in a secured environment if they face difficulties or possible negative effects of the intervention. The content of the program is based on an already established internet-based self-help program against insomnia that was already tested in a previous study.
- CAU (control group): Participants of this arm will get a treatment prescribed by a consulting doctor (care as usual - CAU). After the 2-month course participants will pass the post-treatment assessment followed by the 3-month follow-up and post-follow-up assessment. Then provided completion of all the assessments and satisfying eligibility criteria participants of this arm will get the access to the 2-month iCBT-I course followed by the post-treatment assessment
  internet-delivered cognitive-behavioral therapy for insomnia (iCBT-I): The 2-month intervention consists of educational material divided into 8 modules, which provide the rationale for the CBT-I interventions: sleep restriction; stimulus control; cognitive techniques; relaxation techniques. Information is presented in 10-minute videolectures.
  The program includes a sleep diary to insert bedtime and waketime, sleep latency, total sleep time, night awakenings.
  All material will be delivered through the internet program and expected to be elaborated by the patient but with the opportunity to contact a specialist via the feedback form (guidance on request) in a secured environment if they face difficulties or possible negative effects of the intervention. The content of the program is based on an already established internet-based self-help program against insomnia that was already tested in a previous study.
  Care as usual (CAU): Intervention includes all variety of therapy methods that can be prescribed by medical doctors (MD)
Arm/Group | iCBT-I + CAU | CAU (control group)
Number analyzed (Participants) | 53 | 1
score on a scale | 32.8 (25.1) | 10 (NA) — Below the level of detection Only 1 participant of CAU group has answered this question

20. Secondary Outcome: Number of Completed Modules
Description: Measure of adherence. Program-derived outcome measuring, how many modules were completed (i.e. videolecture, answers to the questions after videolecture)
Time Frame: as for outcome 18
Measure: Mean (Standard Error); unit: number of completed modules
Groups:
- CAU group: Care as usual (CAU): Intervention includes all variety of therapy methods that can be prescribed by medical doctors (MD): pharmacotherapy, behavioral recommendations, face-to-face psychotherapy. Prescriptions may be made during the first visit to MD, or at any point in the study on a next doctor visit, or during visits to the doctors of other medical centers.
Arm/Group | iCBT-I + CAU | CAU group
Number analyzed (Participants) | 53 | 54
number of completed modules | 6.54 (2.41) | 4.93 (3.28)

21. Secondary Outcome: Total Time Spent on the iCBT-I Website
Description: measure of adherence. Program-derived outcome
Time Frame: as for outcome 18
Population: although data were automatically collected by the software, its further analysis was not possible due to the technical problems to extract the data and to use them in the analysis, since it could be done only by a software developer who has left the project earlier. Data are not planned to be analyzed in the future
Measure: Mean (Standard Error); unit: minutes
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Time Spent on Each Module
Description: measure of adherence. Program-derived outcome
Time Frame: as for outcome 18
Population: as for outcome 21
Measure: Mean (Standard Error); unit: minutes
Arm/Group | iCBT-I + CAU | CAU (control group)
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Number of Completed Sleep Diaries
Description: measure of adherence. Program-derived outcome
Time Frame: as for outcome 18
Measure: Mean (Standard Error); unit: number of completed modules
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
number of completed modules | 6.54 (2.41) | 4.93 (3.28)

24. Secondary Outcome: Usage of the Support
Description: number of referrals to the supporting psychologist through the feedback form. Program-derived outcome
Time Frame: as for outcome 18
Measure: Mean (Standard Error); unit: number of emails to the support
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
number of emails to the support | 9.44 (4.14) | 7.74 (4.03)

25. Secondary Outcome: Attention Seeking From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Attention seeking is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 2.24 (0.89) | 2.04 (0.77)

26. Secondary Outcome: Callousness From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Callousness is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ICBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.26 (0.37) | 1.33 (0.44)

27. Secondary Outcome: Deceitfulness From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Deceitfulness is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ICBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.49 (0.48) | 1.57 (0.45)

28. Secondary Outcome: Depressivity From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Depressivity is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.23 (0.34) | 1.43 (0.44)

29. Secondary Outcome: Distractability From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Distractability is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 2.10 (0.73) | 2.27 (0.77)

30. Secondary Outcome: Eccentricity From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Eccentricity is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.67 (0.80) | 1.62 (0.71)

31. Secondary Outcome: Emotional Lability From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Emotional lability is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.70 (0.65) | 1.79 (0.53)

32. Secondary Outcome: Grandiosity From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Grandiosity is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.65 (0.59) | 1.56 (0.56)

33. Secondary Outcome: Hostility From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Hostility is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.75 (0.65) | 2.01 (0.55)

34. Secondary Outcome: Impulsivity From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Impulsivity is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.69 (0.64) | 1.63 (0.57)

35. Secondary Outcome: Intimacy Avoidance From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Intimacy avoidance is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.70 (0.76) | 1.82 (0.68)

36. Secondary Outcome: Irresponsibility From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Irresponsibility is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.34 (0.36) | 1.35 (0.40)

37. Secondary Outcome: Manipulativeness From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Manipulativeness is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.65 (0.52) | 1.65 (0.52)

38. Secondary Outcome: Perceptual Dysregulation From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Perceptual dysregulation is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.16 (0.34) | 1.14 (0.27)

39. Secondary Outcome: Perseveration From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Perseveration is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 2.08 (0.68) | 2.24 (0.65)

40. Secondary Outcome: Restricted Affectivity From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Restricted affectivity is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.91 (0.56) | 2.13 (0.57)

41. Secondary Outcome: Rigid Perfectionism From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Rigid perfectionism is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 2.21 (0.61) | 2.28 (0.72)

42. Secondary Outcome: Risk Taking From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Risk taking is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.50 (0.56) | 1.52 (0.65)

43. Secondary Outcome: Separation Insecurity From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Separation insecurity is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 2.24 (0.70) | 2.49 (0.69)

44. Secondary Outcome: Submissiveness From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Submissiveness is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 2.17 (0.72) | 2.16 (0.64)

45. Secondary Outcome: Suspiciousness From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Suspiciousness is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.58 (0.56) | 1.57 (0.54)

46. Secondary Outcome: Unusual Beliefs Experience From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Unusual beliefs experience is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.24 (0.36) | 1.13 (0.22)

47. Secondary Outcome: Withdrawal From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Withdrawal is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.81 (0.68) | 2.08 (0.65)

48. Secondary Outcome: Anhedonia From Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Predictive Effect on ISI Improvement
Description: 100-item self-report inventory designed to assess the 25 pathological personality trait facets and the 5 domains based on the dimensional trait model (DSM-5 Section III). Anhedonia is one of the personality trait facets and its total score is a sum of 4 items which are rated on a 4-point Likert scale from 0 (very false or often false) to 3 (very true or often true). Therefore the total score may vary from 0 to 12, where higher value represent the higher expression of this pathological facet
Time Frame: Once at baseline assessment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | iCBT-I + CAU | Care as usual (CAU)
Number analyzed (Participants) | 53 | 54
units on a scale | 1.69 (0.59) | 1.89 (0.54)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | iCBT-I + CAU | Care as Usual (CAU)
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/54
Other Adverse Events (participants affected / at risk) | 0/53 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT04300218/Prot_SAP_000.pdf